CLINICAL TRIAL: NCT06938399
Title: Motiva Implants® Post-Approval Study (PAS) Protocol for Motiva SmoothSilk® Round Ergonomix® ('Ergonomix®') and SmoothSilk® Round ('Round') Breast Implants in Subjects Who Are Undergoing Primary Breast Augmentation, Revision Augmentation and Other Aesthetic Procedures
Brief Title: Motiva Implants® Post-Approval Study
Acronym: Motiva PAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Motiva USA LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001005; P230005 (Other: FDA)
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Breast Implant
Keywords: Breast Implants; Breast Surgery; Breast Augmentation; Breast Revision; Silicone Implants

STUDY DESIGN:
Intervention Model Description: Multicenter, 3 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Primary Augmentation (Other): Subjects age 22 and over, indicated to increase breast size
  Interventions: Device: Silicone gel-filled breast implants - Motiva Implants®
- Revision Augmentation (Other): Revision surgery to correct or improve the results of a previous breast augmentation
  Interventions: Device: Silicone gel-filled breast implants - Motiva Implants®
- Control Group (Other): Aesthetic procedure other than breast implant surgery
  Interventions: Other: Aesthetic Surgery

INTERVENTIONS:
Device: Silicone gel-filled breast implants - Motiva Implants® — Breast Surgery
  Other Names: Breast Augmentation
  Arms: Primary Augmentation; Revision Augmentation
Other: Aesthetic Surgery — Aesthetic procedure other than breast implant surgery
  Other Names: Aesthetic procedure
  Arms: Control Group

SUMMARY:
This study examines the general post-market use and safety of Motiva Implants® and gathers and assesses selected safety and effectiveness data about their post market performance and experience.

DETAILED DESCRIPTION:
Prospective, non-randomized, multicenter study including baseline (preoperative), operative, and postoperative data collection annually Years 1-10.

ELIGIBILITY:
Inclusion Criteria Motiva Implants®:

* Female
* Patient is seeking one of the following procedures: -Primary Breast Augmentation: age 22 and over, indicated to increase breast size -Revision Breast Augmentation: removal and replacement of breast implants (revision) to correct or improve the results of a previous breast augmentation
* Patient has adequate tissue available to cover implant(s)
* Willingness to follow all study requirements
* Signs an Informed Consent
* Agrees to have device returned to the Sponsor, if explanted
* Willing to undergo Computed Tomography Scan (CT), ultrasound, or MRI evaluation, if medically advised

Inclusion Criteria Control group:

* Is 22 years of age or older
* Female
* Is a candidate for aesthetic surgery (such as liposuction, rhinoplasty, face-lift)
* Signs an Informed Consent
* Willingness to follow all study requirements

Exclusion Criteria Motiva Implants®:

* Has any breast disease considered to be pre-malignant in one or both breasts or is reporting mutations in BRCA1 or BRCA2
* Has inadequate or unsuitable tissue (e.g., due to radiation damage, ulceration, compromised vascularity, history of compromised wound healing)
* Has an active infection anywhere in their body
* Is pregnant or nursing, or has had a full-term pregnancy or lactated within 6 months of enrollment
* Is taking any drugs that would interfere with blood clotting, or that might result in elevated risk and/or significant postoperative complications
* Has any medical condition such as obesity (BMI >40), diabetes, autoimmune disease, chronic lung or severe cardiovascular disease that might result in unduly high surgical risk and/or significant postoperative complications
* Has any connective tissue/autoimmune disorder or rheumatoid disease, such as systemic lupus erythematosus, discoid lupus, scleroderma, or rheumatoid arthritis, among others
* Has a history of psychological characteristics that are unrealistic or unreasonable given the risks involved with the surgical procedure
* Has been implanted with any non-FDA approved breast implant
* Has been implanted with any silicone implant other than breast implants
* HIV positive (based on medical history)
* Has been diagnosed with Breast Implant Associated-Anaplastic Large Cell Lymphoma (BIA-ALCL)

Exclusion Criteria Control group:

* Has a history of silicone implants (anywhere in the body)
* Plans to undergo silicone breast implant surgery during the course of the study
* Has an active infection anywhere in their body
* Has a history of cancer (except skin cancer)
* Is taking any drugs that would interfere with blood clotting, or that might result in elevated risk and/or significant postoperative complications
* Has any medical condition such as obesity (BMI >40), diabetes, autoimmune disease, chronic lung or severe cardiovascular disease that might result in unduly high surgical risk and/or significant postoperative complications
* Has any connective tissue/autoimmune disorder or rheumatoid disease, such as systemic lupus erythematosus, discoid lupus, scleroderma, or rheumatoid arthritis, among others

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2037-04-01 (Estimated); Study Completion 2037-07-31 (Estimated)

PRIMARY OUTCOMES:
Investigate the incidence of connective tissue disease (CTD) signs and symptoms in Motiva implanted participants compared to the incidence in control participants | 10 Years
  Analysis of Patient-Reported incidence of Connective Tissue Diseases (CTDs) and related systemic symptoms, collected through a questionnaire that includes the PROMIS-29 Survey

SECONDARY OUTCOMES:
Investigate the incidence of Reproductive Complications, Cancer Diagnoses, Local Complications in Motiva implanted participants compared to the incidence in control participants, where data collection allows; and investigate patient satisfaction | 10 Years
  Analysis of Patient-Reported safety and satisfaction collected through a Follow-Up Questionnaire and 5-point Likert scale
Assess the impact of RFID on imaging | 10 Years
  Frequency of imaging impact among participants implanted with devices containing RFID

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - J. Gerald Minniti, M.D., F.A.C.S., Beverly Hills, California
  - AESTHETX Center, Camp Pendleton, California
  - Align Surgical Associates Inc, San Francisco, California
  - Schwartz Aesthetic Institute, Westlake Village, California
  - The Center for Cosmetic Surgery, Denver, Colorado
  - Advanced Plastic Surgery, LLC, Washington D.C., District of Columbia
  - Careaga Plastic Surgery, Coral Gables, Florida
  - Renee Burke Plastic Surgery, Aesthetics, & Med Spa, South Barrington, Illinois
  - CaloAesthetics® Plastic Surgery Center, Louisville, Kentucky
  - The Wall Center for Plastic Surgery, Shreveport, Louisiana
  - Center for Plastic Surgery, Chevy Chase, Maryland
  - Parkcrest Plastic Surgery, St Louis, Missouri
  - Delaware Valley Plastic Surgery, Cherry Hill, New Jersey
  - Caroline A. Glicksman MD, Sea Girt, New Jersey
  - Mark D. Epstein, MD, FACS Center for Aesthetic Surgery, Hauppauge, New York
  - Neinstein Plastic Surgery, New York, New York
  - HKB Cosmetic Surgery, Charlotte, North Carolina
  - Capizzi, MD Cosmetic Surgery & Med Spa, Charlotte, North Carolina
  - Restora Austin Plastic Surgery Center, Austin, Texas
  - Austin Plastic Surgeon, Austin, Texas
  - Southwest Plastic Surgery, El Paso, Texas
  - Kristy Hamilton MD, FACS, Houston, Texas
  - North Texas Plastic Surgery, Southlake, Texas
  - The Plastics Clinic & SPA, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teuwen MMH, Knaapen IRE, Vliet Vlieland TPM, Schoones JW, van den Ende CHM, van Weely SFE, Gademan MGJ. The use of PROMIS measures in clinical studies in patients with inflammatory arthritis: a systematic review. Qual Life Res. 2023 Oct;32(10):2731-2749. doi: 10.1007/s11136-023-03422-0. Epub 2023 Apr 27. PMID 37103773
- [Background] Sun K, Eudy AM, Harris N, Pisetsky DS, Criscione-Schreiber LG, Sadun RE, Doss J, Clowse MEB, Rogers JL. Using PROMIS-29 to determine symptom burdens in the context of the Type 1 and 2 systemic lupus erythematosus (SLE) model: a cross sectional study. J Patient Rep Outcomes. 2023 Dec 21;7(1):136. doi: 10.1186/s41687-023-00678-5. PMID 38127169
- [Background] Hinchcliff ME, Beaumont JL, Carns MA, Podlusky S, Thavarajah K, Varga J, Cella D, Chang RW. Longitudinal evaluation of PROMIS-29 and FACIT-dyspnea short forms in systemic sclerosis. J Rheumatol. 2015 Jan;42(1):64-72. doi: 10.3899/jrheum.140143. Epub 2014 Nov 1. PMID 25362656
- [Background] Bingham Iii CO, Gutierrez AK, Butanis A, Bykerk VP, Curtis JR, Leong A, Lyddiatt A, Nowell WB, Orbai AM, Bartlett SJ. PROMIS Fatigue short forms are reliable and valid in adults with rheumatoid arthritis. J Patient Rep Outcomes. 2019 Feb 21;3(1):14. doi: 10.1186/s41687-019-0105-6. PMID 30790155
- [Background] Bartlett SJ, Gutierrez AK, Andersen KM, Bykerk VP, Curtis JR, Haque UJ, Orbai AM, Jones MR, Bingham CO 3rd. Identifying Minimal and Meaningful Change in a Patient-Reported Outcomes Measurement Information System for Rheumatoid Arthritis: Use of Multiple Methods and Perspectives. Arthritis Care Res (Hoboken). 2022 Apr;74(4):588-597. doi: 10.1002/acr.24501. Epub 2022 Mar 3. PMID 33166066
- [Background] Almalag HM, Almaghlouth I, Dabbagh R, Alsalem AR, Alrajban FN, Algarni SA, Alosaimi FN, Alassaf MI, Alshamrani MA, Alzomia S, Alanazi B, Alalwan T, Alkhalaf A, Bedaiwi M, Omair MA. Prevalence of fatigue functional and social impairment among patients with rheumatic diseases compared to patients without: A cross-sectional comparison. Medicine (Baltimore). 2023 Mar 3;102(9):e33151. doi: 10.1097/MD.0000000000033151. PMID 36862854